CLINICAL TRIAL: NCT01103661
Title: Feasibility Study For Safety and Efficacy Evaluation Of The Combined Ablation Procedure For The Treatment Of LongStanding Persistent Atrial Fibrillation
Brief Title: Safety and Efficacy Study of The Combined Ablation Procedure To Treat Longstanding Persistent Atrial Fibrillation
Acronym: CAPstopsLSPAF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: nContact Surgical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAL-1140
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2013-04

CONDITIONS: Atrial Fibrillation
Keywords: Longstanding Persistent Atrial Fibrillation; AF; Chronic AF; RF Ablation; nContact Surgical; Therapy Cool Path Ablation Catheter; St. Jude Medical
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Numeris-AF Guided Coagulation System (Other)
  Interventions: Device: Numeris®-AF Guided Coagulation System with VisiTrax®

INTERVENTIONS:
Device: Numeris®-AF Guided Coagulation System with VisiTrax® — Combined epicardial / endocardial procedure using the nContact Numeris®-AF Guided Coagulation System with VisiTrax® epicardially and the St. Jude Medical Therapy™ Cool Path™ Ablation Catheter endocardially.

SUMMARY:
This is a multi-center, prospective open label, feasibility study evaluating the safety and efficacy of the combined ablation procedure for the treatment of longstanding persistent atrial fibrillation.

DETAILED DESCRIPTION:
The purpose of this feasibility study is to evaluate the safety and efficacy of the epicardial / endocardial combined procedure using the nContact Numeris®-AF Guided Coagulation System with VisiTrax® epicardially and the St. Jude Medical Therapy™ Cool Path™ Ablation Catheter endocardially to treat longstanding persistent Atrial Fibrillation (AF) patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years; < 80 years
* Left atrium less than or equal to 6.5 cm (TTE)
* History of AF for less than or equal to 10 years
* Provided written informed consent
* Symptomatic longstanding persistent Atrial Fibrillation (AF).

Exclusion Criteria:

* Patients requiring concomitant surgery
* Left ventricular ejection fraction < 30%
* Pregnant or planning to become pregnant during study
* Co-morbid medical conditions that limit one year life expectancy
* Measured left ventricular wall thickness > 1.5 cm
* History of coagulopathy
* Previous cardiac surgery
* History of pericarditis
* Previous cerebrovascular accident (CVA), excluding fully resolved TIA
* Patients who have active infection or sepsis
* Patients who have uncorrected reversible cause(s) of AF
* Patients who are contraindicated for anticoagulants
* Patients who are being treated for arrhythmias other than AF
* Patients who have had any previous AF or left atrial catheter ablation
* Current participation in another clinical investigation of a medical device or a drug, or recent participation in such a study within 30 days prior to study enrollment
* Not competent to legally represent him or herself (e.g., requires a guardian or caretaker as a legal representative).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-04; Primary Completion 2012-10 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
AF free, off all Class I and III Anti Arrhythmic Drugs (AADs) | 12 months
  The primary efficacy data will be an evaluation of the number of subjects free from AF and free of all Class I and III Anti Arrhythmic Drugs (AADs) from 3 months through 12 months post procedure.

SECONDARY OUTCOMES:
AF free regardless of the Class I and III AADs status | 12 months
  The secondary efficacy data will be an assessment of the number of subjects free from AF regardless of their Class I and III AADs status from 3 months through 12 months post procedure.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - The Care Group, St Vincent Hospital, Indianapolis, Indiana
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Texas Cardiac Arrhythmia Institute, St. David's Hospital, Austin, Texas
  - Cardiothoracic Surgical Associates, CJW Medical Center, Richmond, Virginia